CLINICAL TRIAL: NCT04518917
Title: Sing for Your Saunter: Using Self-generated Rhythmic Cues to Enhance Gait in Parkinson's - Dementia Supplement
Brief Title: Sing for Your Saunter - Dementia Supplement
Acronym: SFYS-D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Gammon M Earhart, Director, Program in Physical Therapy, Washington University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AT010753-02S1
Record Dates: First submitted 2020-08-15; First posted 2020-08-19 (Actual); Results first posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-11

CONDITIONS: Parkinson Disease; Parkinson Disease Dementia
Keywords: Parkinson disease; Music; Mental singing; Gait
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Parkinson disease plus dementia (Other): Participants will have a diagnosis of Parkinson disease plus dementia.
  Interventions: Behavioral: Mentally Singing; Behavioral: Listening to music

INTERVENTIONS:
Behavioral: Mentally Singing — Participants sing their song in their head and match their footfalls to the beat.
Behavioral: Listening to music — Participants listen to their song and match their footfalls to the beat.

SUMMARY:
Older adults, and particularly those with Parkinson disease (PD), may experience walking difficulties that negatively impact their daily function and quality of life. People that have PD plus dementia are also likely to experience walking difficulties. This project will examine the impact of music and mentally singing on walking performance, with a goal of understanding what types of rhythmic cues are most helpful. Pilot work from the investigators suggests that imagined, mental singing (i.e., singing in head) while while walking helps people walk faster with greater stability, whereas walking to music also helps people walk faster but with reduced stability.

In this study, the investigators will recruit people who have PD plus dementia. The investigators will compare walking while mentally singing and walking while listening to music, using personalized cues tailored to each person's walking performance. The investigators hypothesize temporal variability of gait will be lower in the mental singing and singing conditions compared to listening to music; and that mental singing, singing, and listening to music will elicit similar improvements in stride length.

DETAILED DESCRIPTION:
During this observational study, participants will attend one visit in the laboratory. The visit will include participants wearing wearable sensors during the following tasks: walking with no cues (UNCUED), walking while listening to music (MUSIC), and walking while mentally singing (MENTAL SINGING). The wearable sensors will measure gait parameters including gait speed, stride length, and stride time variability.

ELIGIBILITY:
Inclusion Criteria:

* at least 30 years of age
* diagnosis of idiopathic, typical Parkinson disease according to the UK Brain Bank Criteria
* Hoehn & Yahr stages 2-3 (mild to moderate disease severity)
* normal or corrected hearing
* stable on all PD medications for at least 2 months prior to study entry
* dementia as defined by a Clinical Dementia Rating (CDR) score of 0.5-1.0 (very mild to mild dementia)
* score of ≥ 1 on the MDS-UPDRS-III Item #10 indicating observable gait impairment
* a score of 1 or less on item #7 on the freezing of gait questionnaire
* able to walk for 10 continuous minutes independently

Exclusion Criteria:

* diagnosis of any other neurological condition
* unstable medical or concomitant illnesses or psychiatric conditions which, in the opinion of the investigators, would preclude successful participation
* cardiac problems that interfere with ability to safely participate (i.e., uncontrolled congestive heart failure, myocardial infarction in past 6 months, complex cardiac arrhythmias, significant left ventricular dysfunction, dyspnea on exertion, chest pain or pressure, resting tachycardia (>100 beats/min); uncontrolled BP (resting systolic BP >160 mmHg or diastolic BP >100 mmHg))
* orthopedic problems in the lower extremities or spine that may limit walking (i.e., severe arthritis, spinal stenosis)
* uncontrolled tremor or dyskinesia while on PD medications

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gammon Earhart, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine Program in Physical Therapy, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Parkinson Disease Plus Dementia
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Parkinson Disease Plus Dementia: Participants will have a diagnosis of Parkinson disease plus dementia.
  Mentally Singing: Participants sing their song in their head and match their footfalls to the beat.
  Listening to music: Participants listen to their song and match their footfalls to the beat.
  Singing: Participants will sing their song out loud and match their footfalls to the beat.
Arm/Group | Parkinson Disease Plus Dementia
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.7 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Velocity
Description: Measured with wearable sensors by APDM Wearable Technology
Time Frame: Baseline
Population: For the uncued column the condition is by definition one with no cues. As such, there are no data for the 90, 100, 110, and 120% cue rows as these are only relevant for the cued conditions. Similarly, the mental singing and music conditions are by definition cued so there are no data for the no cue row as that is only relevant for the uncued condition.
Measure: Mean (Standard Deviation); unit: meters per second
Groups:
- Mental Singing: Mentally Singing: Participants sing their song in their head and match their footfalls to the beat.
- Music: Listening to music: Participants listen to their song and match their footfalls to the beat.
- Uncued: Participants walking without any cues (i.e., no music, no singing)
Arm/Group | Mental Singing | Music | Uncued
Number analyzed (Participants) | 17 | 17 | 17
meters per second
  90% tempo cue: number analyzed (Participants) | 17 | 17 | 0
  90% tempo cue | .977 (.234) | .960 (.243) |
  100% tempo cue: number analyzed (Participants) | 17 | 17 | 0
  100% tempo cue | 1.042 (.27) | 1.011 (.255) |
  110% tempo cue: number analyzed (Participants) | 17 | 17 | 0
  110% tempo cue | 1.070 (.286) | 1.072 (.279) |
  120% tempo cue: number analyzed (Participants) | 17 | 17 | 0
  120% tempo cue | 1.083 (.29) | 1.072 (.301) |
  No cue: number analyzed (Participants) | 0 | 0 | 17
  No cue |  |  | 1.02 (0.04)

2. Primary Outcome: Stride Length
Description: Measured with wearable sensors by APDM Wearable Technology
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: meters
Groups:
- Uncued: Walking without any cues (i.e., no music, no singing)
Arm/Group | Mental Singing | Music | Uncued
Number analyzed (Participants) | 17 | 17 | 17
meters
  90% cue tempo: number analyzed (Participants) | 17 | 17 | 0
  90% cue tempo | 1.085 (.254) | 1.089 (.260) |
  100% cue tempo: number analyzed (Participants) | 17 | 17 | 0
  100% cue tempo | 1.116 (.262) | 1.103 (.258) |
  110% cue tempo: number analyzed (Participants) | 17 | 17 | 0
  110% cue tempo | 1.130 (.274) | 1.130 (.266) |
  120% cue tempo: number analyzed (Participants) | 17 | 17 | 0
  120% cue tempo | 1.128 (.265) | 1.129 (.272) |
  No cue: number analyzed (Participants) | 0 | 0 | 17
  No cue |  |  | 1.12 (0.03)

ADVERSE EVENTS:
Time Frame: During single lab visit that took a few hours
Description: Monitoring in real time during single session during which participants were continually supervised
Arm/Group | Parkinson Disease Plus Dementia
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-15): https://cdn.clinicaltrials.gov/large-docs/17/NCT04518917/Prot_SAP_000.pdf